CLINICAL TRIAL: NCT04138342
Title: Fluorescent Nanoparticles Conjugated Long-acting Somatostatin Analog for Potent Suppression and Bioimaging Breast Cancer
Brief Title: Topical Fluorescent Nanoparticles Conjugated Somatostatin Analog for Suppression and Bioimaging Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed A. H. Abdellatif, Associate Professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Qassim QDs-VELD
Record Dates: First submitted 2019-10-07; First posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer; Skin Cancer; Skin Diseases
MeSH Terms: conditions — Breast Neoplasms; Skin Neoplasms; Skin Diseases | interventions — Floderm topical cream

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quantum dots nanoparticles group (Active Comparator): A group of female volunteers infected with breast cancer will receive topical Quantum dots in different dosage forms.
  Interventions: Drug: Quantum dots coated with veldoreotide
- Topical approved placebo cream (Placebo Comparator): A group of female volunteers infected with breast cancer will receive placebo cream as a negative control.
  Interventions: Drug: Topical approved placebo

INTERVENTIONS:
Drug: Quantum dots coated with veldoreotide — The active group will receive Quantum dots coated with veldoreotide in different topical dosage forms as an anti-cancer drug.
  Other Names: Topical cream
  Arms: Quantum dots nanoparticles group
Drug: Topical approved placebo — The placebo group will receive topical FDA approved in different dosage forms as a negative control drug.
  Other Names: Topical placebo gel or cream
  Arms: Topical approved placebo cream

SUMMARY:
Breast cancer is a communal malignant disease between Saudi females, with a popularity of 21.8%. Since binding to somatostatin receptors (SSTR) induces no immunogenicity in vivo, somatostatin analog (veldoreotide) (VELD) may be suitable for delivering anti-cancer drugs to target and bioimaging the cancer cells. This work aimed to deliver CdS/ZnS core-shell type quantum dots with carboxylic acid-functionalized (QDs-COOH) which is bioimaging and anticancer nanoparticles decorated VELD as SSTR agonist with anti-cancer activity in the form of topical cream to be deposited deep in the breast periphery.

DETAILED DESCRIPTION:
QDs-COOH will be conjugated to the N terminal of phenylalanine of VELD when the reaction proceeded at pH 7. Topical cream will be adapted to deliver the conjugated system for maximum deposition through breast cancer cells using emulsion technology. The formulated nanoparticles and cream will be characterized for size using dynamic light scattering, drug-polymer interaction using FTIR, and morphology using SEM. Cellular uptake, permeability and cell viability study of the successful system of interest will be studied in cell culture models using different breast cell lines. Moreover, the in vivo study will also proceed on rats induced breast cancer. Finally, the nanoparticles loaded in a topical cream will be applied with clinical trial approvement on the human breast cancer for bioimaging and treating breast cancer. This work is to present a novel formulation for treatment and bioimaging of breast cancer which can deliver safely to the patients in a high dose to the affected tumor cells.

ELIGIBILITY:
Inclusion Criteria:

1. Women, 25 to 60 years old.
2. Breast biopsy within 60 days of registration (dosing) without proof of aggressive cancer in any specimen;
3. Invasive breast cancer verified by histology of ER ≥ 10% (all test results should be checked and validated by the Pathology Department of the involved institution);
4. Participants performed traditional regional radical therapy (modified or moderate radical mastectomy) with or without neoadjuvant/adjuvant chemotherapy or radiotherapy;
5. Hemoglobin ≥ 90 g / L, neutrophils ≥ 1.5 × 109/L, platelets ≥ 75 × 109/L, AST and ALT ≤ 2.5 times the upper limit for natural (ULN), creatinine serum and urea nitrogen ≤ ULN.

Exclusion Criteria:

1. Patients have previously received any other treatment or have begun adjuvant therapy.
2. There are any comorbidities that may increase the level of sex hormones: pituitary adenomas, ovarian cancers, thymic carcinomas, etc.
3. There are any comorbidities that may decrease sex hormone rates such as hyperthyroidism, hypothyroidism, cirrhosis, extreme obesity, Turner syndrome, lack of sex hormone synthetase, intracranial tumors, pituitary atrophy, etc. Patients have undergone and expected suppression of ovariectomy and ovarian activity.
4. Patients have been diagnosed with other test drugs for the next 2 months.
5. People of child-bearing age who are not willing to take effective contraception through therapy. Serious non-maligned tumor comorbidities can impair long-term follow-up.
6. Patients have a family history of endometrial, reproductive or other gynecological malignancies. Transvaginal testing indicated more severe ovary defects and endometrial thickening.
7. Patients had thrombotic incidents such as a cerebrovascular injury (including a transient ischemic attack), deep venous thrombosis, and pulmonary embolism within 6 months of the start of the research.
8. Serious insufficiency of the liver with Child-Pugh C class. Serious heart disease of New York Heart Association (NYHA) class ≥III. Patients are considered to be severely allergic to medications.
9. Patients have a record of other malignancies over the last five years, with the exception of cutaneous basal cell carcinoma and cervical in situ carcinoma that has been healed. In other instances, investigators do not feel the topics are acceptable for study participants.
10. Pregnant or lactating women (women of childbearing age should receive a negative pregnancy test within 14 days of the first dosage or, if pregnant, clinicians are required to undergo an ultrasound review to exclude childbirth).

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-06-14 (Estimated); Study Completion 2022-12-13 (Estimated)

PRIMARY OUTCOMES:
Growth inhibition was measured using the sulforhodamine B-based assay. | 6 months
  QDs-VELD have anticancer activity. This study will be determined by measuring the growth inhibition of anticancer activity for QDs-VELD.
Amount of QDs-VELD fluorescent QDs-VELD in the breast periphery due to the fluorescence of QDs using flow cytometry. | 6 months
  The bioimaging effect for scintigraphy of breast cancer.
Growth inhibition was measured by visual determination of breast cancer cells. | 6 months
  QDs-VELD have anticancer activity. This study will be determined by measuring the growth inhibition of anticancer activity for QDs-VELD.

SECONDARY OUTCOMES:
Stable topical quantum dots coated veldoreotide | three months
  Stability test will be studied for dosage forms. The test will carried out by standing the products on shelf life for three months. The stability test will be recorded using high performance liquid chromatography each thee days.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed AH Abdellatif, PhD, Principal Investigator — Qassim University
Locations (4):
- Assiut Clinic, Asyut, Egypt
- Saudi Arabia (3):
  - Buraidah Clinic, Buraidah, Al Qassim
  - Faculty of Pharmacy, Buraidah, Al-Qassim Region
  - Pharmaceutics dept., Faculty of Pharmacy, Qassim University, Buraidah, Al-Qassim Region

IPD SHARING:
Plan to Share IPD: No
The authors could not decide until now a plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Result] Clive S, Gardiner J, Leonard RC. Miltefosine as a topical treatment for cutaneous metastases in breast carcinoma. Cancer Chemother Pharmacol. 1999;44 Suppl:S29-30. doi: 10.1007/s002800051114. PMID 10602908
- [Result] Doroshow JH. Redox modulation of chemotherapy-induced tumor cell killing and normal tissue toxicity. J Natl Cancer Inst. 2006 Feb 15;98(4):223-5. doi: 10.1093/jnci/djj065. No abstract available. PMID 16478735